CLINICAL TRIAL: NCT00630578
Title: Improving Effectiveness: Treatment Outcome Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Trauma Recovery, St Louis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Tara Galovski, University of Missouri- St. Louis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH074937-01A2 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic Stress Disorder; Physical Assault; Physical Abuse; Sexual Assault; Sexual Abuse; Interpersonal Assault; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cognitive Processing Therapy
  Interventions: Behavioral: Cognitive Processing Therapy
- 2 (No Intervention): Arm 2 participants will monitor their symptoms for a period of 10 weeks, prior to being crossed over into active treatment. This will allow investigators to account for the passage of time without intervention when tracking symptoms.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Clients will receive between 4 and 20 sessions of Cognitive Processing Therapy.

SUMMARY:
This proposal seeks to increase the effectiveness of an existing treatment strategy, cognitive processing therapy (CPT), for the remediation of Posttraumatic Stress Disorder among crime victims by varying the duration and content of the intervention in accordance with participants' needs. A secondary goal is to identify predictors of duration of treatment necessary to achieve good end state functioning, including individual and trauma variables, cognitive and emotional variables, and Axis II pathology. Finally, by including a sample of male participants, the generalizability of CPT will be tested. It is anticipated that these modifications will speed the dissemination of CPT to community practice thus benefiting more trauma victims. Fifty subjects will be randomly assigned to either the modified CPT condition or to a symptom-monitoring, minimal attention condition designed to control for the effects of the daily monitoring and the passage of time. Utilizing a semicrossover design, the control condition will be crossed over to the active treatment, allowing for a replication within the study. The entire treated sample (N = 50) will be compared to a sample (N = 50) receiving strict 12-session protocol-driven CPT through the course of a recent study conducted at the same site using the same primary outcome measures. Conducting the proposed study will have important implications on advancing the ecological validity and effectiveness of applied research on PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be survivors of interpersonal assault, who are at least three months post-crime at the time of their participation and who meet criteria for a diagnosis of PTSD. There is no upper time limit on time since crime for participation.

Exclusion Criteria:

* Exclusion criteria for participants include psychosis, mental retardation, active suicidality, parasuicidality, or current addiction to drugs or alcohol. In the case of apparent illiteracy, we will try to accommodate the individual as much as possible to maximize success in the program. In addition, participants cannot be in a currently abusive relationship or being stalked. For marital rape or domestic violence, the participant must have been out of the relationship for at least three months. Participants may continue the use of any medications throughout the study. However, participants must be willing to keep the medication usage stable for the duration of the study and must be stabilized on any new medication for one month prior to initial assessment. Participants will sign a contract to this effect. All medication use will be tracked throughout the course of the study on the daily symptom monitoring diaries, including over the counter medications. Finally, participants can have received any therapy in the past with the exception of CPT. They may be receiving concurrent therapy as long as it is not trauma-focused. Allowing subjects to continue with concurrent therapy offers them the option to continue with established supports and more closely mimics clinical practice and the generalizability of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Good end-state functioning: Beck Depression Inventory-II and Posttraumatic Distress Scale Scores | 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tara Galovski, PhD, Principal Investigator — Center for Trauma Recovery, University of Missouri- St. Louis
Locations (1):
- Center for Trauma Recovery, St Louis, Missouri, United States

REFERENCES:
- [Derived] Alpert E, Carpenter JK, Smith BN, Woolley MG, Raterman C, Farmer CC, Kehle-Forbes SM, Galovski TE. Leveraging observational data to identify in-session patient and therapist predictors of cognitive processing therapy response and completion. J Trauma Stress. 2023 Apr;36(2):397-408. doi: 10.1002/jts.22924. Epub 2023 Mar 29. PMID 36987703